CLINICAL TRIAL: NCT01489735
Title: Observational Non-interventional Study on the Use of International GerdQ Questionnaire for the Diagnosis of Gastroesophageal Reflux Disease in the Russian Practice
Brief Title: The Use of International GerdQ Questionnaire
Acronym: GERDq
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GRU-XXX-2011/1
Record Dates: First submitted 2011-12-02; First posted 2011-12-12 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; GERD Q QUESTIONNAIRE
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
There are three main directions for use GerdQ in practice. First of all, GerdQ can be used to diagnose GERD with an accuracy comparable to the accuracy of diagnosis of GERD by the specialist (gastroenterologist). Using GerdQ can evaluate the impact of disease on the patient's life and help in choosing treatment of GERD, as well as direct assessment of treatment efficacy.

In connection with mentioned above, this study is devoted to the estimation of possibility to use GerdQ in routine practice of Russian physicians.

DETAILED DESCRIPTION:
Observational non-interventional study on the use of international GerdQ questionnaire for the diagnosis of gastroesophageal reflux disease in the Russian practice

ELIGIBILITY:
Inclusion Criteria:

* Signing of informed consent to participate in the study
* patients of both sexes, 18 years and older
* planned esophagogastroduodenoscopy

Exclusion Criteria:

* Surgical intervention for upper digestive tract (surgery for gastroesophageal reflux disease, peptic ulcer disease, etc.) In the past
* the presence of contraindications for esophagogastroduodenoscopy or pH-metry
* refusal to sign informed consent
* acceptance of antisecretory drugs (proton pump inhibitors, h2-receptor blockers), antacids and prokinetics for 7 days before enrollment
* Pregnancy
* Confirmed or suspected malignancy
* Impairment of the mental sphere
* Acceptance of nsaids (including acetylsalicylic acid at a dose of 150 mg / day), cytostatics, antibiotics (tetracyclines, lincosamides) at enrollment and during the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLINICAL PRACTICE
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of GerdQ questionnaire = rate of GERD by GerdQ questionnaire (total score ≥8) / number of patients whose GERD was confirmed by instrumental examinations. | Up to 6 months
Specificity of GerdQ questionnaire = rate of GERD by GerdQ questionnaire (total score <8) / number of patients whose GERD diagnosis was excluded on the basis of instrumental examination | Up to 6 months

SECONDARY OUTCOMES:
Sensitivity of GERD diagnosis made by gastroenterologist = result of completion of GerdQ questionnaire / the results of clinical assessment by gastroenterologist. | Up to 6 months
Frequency of GERD diagnosis based on instrumental examination (endoscopy, pH-metry) in studied patients. | Up to 6 months
Prevalence of GERD with the completed GerdQ questionnaire, which corresponds to the proportion (%) of patients with a total score of ≥ 8 in the questionnaire, among study patients. | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Stepanov, Prof, Study Director — AstraZeneca; Vladimir Ivashkin, Prof, Principal Investigator — Head of Inner Disease Department of First Moscow State Medical University named after I.M. Sechenov
Locations (1):
- Research site, Moscow, Russia